CLINICAL TRIAL: NCT01034007
Title: A Pilot Study Investigating the Clinical Use of Tissue Engineered Vascular Grafts in Congenital Heart Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christopher Breuer (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Gunze Limited (Other)
Responsible Party: Sponsor-Investigator, Christopher Breuer, Director of Tissue Engineering, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHIRB12-00357
Record Dates: First submitted 2008-01-29; First posted 2009-12-17 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Single Ventricle Cardiac Anomaly
Keywords: tissue engineered vascular graft
MeSH Terms: interventions — Blood Vessel Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tissue Engineered Vascular Grafts (Experimental)
  Interventions: Combination Product: Tissue Engineered Vascular Grafts

INTERVENTIONS:
Combination Product: Tissue Engineered Vascular Grafts — Patients will undergo EC TCPC interposition grafting with a tissue engineered vascular graft and serial magnetic resonance angiography (MRA)

SUMMARY:
An initial feasibility and safety study evaluating the use of autologous tissue engineered vascular grafts as extra cardiac total cavopulmonary connection (EC TCPC) conduits in children with single ventricle anomalies.

DETAILED DESCRIPTION:
This investigation is a prospective, nonrandomized phase 1 clinical trial determining the safety of the use of tissue engineered vascular grafts as conduits for EC TCPC. Primary end points of the study will include determination of graft failure rates and graft related morbidity and mortality. Graft failure will be defined as any graft narrowing/occlusion or dilation/rupture requiring surgical or endovascular intervention. Graft related morbidity and mortality will include any post-operative complication such as any thromboembolic or infectious event that requires treatment and is thought likely to be caused by the tissue engineered vascular graft as determined by the investigators and confirmed by the data safety monitoring board. All appropriate patients requiring EC TCPC who meet study inclusion/exclusion criteria will be evaluated for enrollment in the clinical trial. After obtaining informed consent from the patient's parents, patients with single ventricle cardiac anomalies will undergo EC TCPC using a tissue engineered conduit. Post-operative care and monitoring will follow an established, standardized, clinical algorithm in which the patient's clinical status including complications and measurements of graft function will be serially evaluated and recorded over a three year period using physical examination, echocardiography, and MRA.

ELIGIBILITY:
Inclusion Criteria:

* single ventricle cardiac anomaly requiring extra cardiac total cavopulmonary connection (EC TCPC).

Exclusion Criteria:

* incomplete inferior vena cava (IVC)

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-12; Primary Completion 2017-12-26 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
graft failure requiring intervention | 3 years

SECONDARY OUTCOMES:
graft growth | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Breuer, MD, Study Chair — Nationwide Children's Hospital, Columbus, Ohio; Toshiharu Shinoka, MD/PhD, Study Chair — Nationwide Children's Hospital, Columbus, Ohio; Mark Galantowicz, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States